CLINICAL TRIAL: NCT01947920
Title: A Randomized, Double-Blind, Placebo-Controlled Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics Following Multiple Ascending Doses of Tramadol Hydrochloride in Healthy Male and Female Subjects
Brief Title: A Dose Ranging Escalation Study of Tramadol Hydrochloride in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Collaborators: Bausch Health Americas, Inc. (Industry); Cipher Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR102458; TRAMPAI1002 (Other: Janssen Scientific Affairs, LLC); V01-TRAA-501 (Other: Valeant Pharmaceuticals International Inc); 2013-01-00 (Other: Cipher Pharmaceuticals Inc)
Record Dates: First submitted 2013-08-13; First posted 2013-09-23 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: Healthy; Pain; Tramadol hydrochloride; Tramadol HCl; Analgesic; QT prolongation; RWJ-26898-002
MeSH Terms: conditions — Pain; Long QT Syndrome | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1: Tramadol HCl 200 mg daily or placebo (Experimental): Participants will receive one capsule of Tramadol hydrochloride (HCl) every 6 hours. Participants assigned to placebo will receive matching placebo capsules. A total of 9 doses will be administered.
  Interventions: Drug: Tramadol HCl, 50 mg; Drug: Placebo
- 2: Tramadol HCl 400 mg daily or placebo (Experimental): Participants will recieve two capsules of Tramadol HCl every 6 hours. Participants assigned to placebo will receive matching placebo capsules. A total of 9 doses will be administered.
  Interventions: Drug: Tramadol HCl, 50 mg; Drug: Placebo
- 3: Tramadol HCl 600 mg daily or placebo (Experimental): Participants will receive three capsules of Tramadol HCl every 6 hours. Participants assigned to placebo will receive matching placebo capsules. A total of 9 doses will be administered.
  Interventions: Drug: Tramadol HCl, 50 mg; Drug: Placebo

INTERVENTIONS:
Drug: Tramadol HCl, 50 mg — 50-mg overencapsulated tablet for oral administration
Drug: Placebo — Size-matching capsules containing an appropriate inactive excipient

SUMMARY:
The purpose of this study is to determine the safety and tolerability profile of tramadol hydrochloride (HCl) given as oral doses every 6 hours, within the range of dosages supported by currently available toxicology and clinical data (200 mg to 600 mg per day).

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), sequential-cohort (time lagged), double-blind (neither the participant or the study doctor will know the name of the assigned treatment), parallel-group, placebo-controlled, 3-arm (participants will be assigned to 1 of 3 treatment groups), single-center, Phase 1 study of multiple ascending doses of tramadol HCl in healthy adult volunteers. Thirty participants (15 men and 15 women) will be sequentially assigned to 1 of 3 treatment groups of 10 subjects each (5 men and 5 women). Participants in each treatment group will receive a total of 9 oral doses (one every 6 hours) of tramadol HCl or placebo, in the ratio of 4:1. The study includes a screening phase and a double-blind treatment phase. The treatment phase will consist of 3 treatment periods separated by a 5-day safety review period before the next ascending dose of study drug is administered to the next group. Participants in each group will be confined to the study center for a total of 5 days, the total duration of each subject's participation will be up to 33 days, including the screening phase. The total duration of the study (completion of all 3 treatment cohorts) will be up-to-approximately 2 months.

ELIGIBILITY:
Inclusion Criteria:

* body mass index between 18 and 30 kg/m², inclusive
* body weight not less than 50 kg
* have a normal electroencephalogram under basic and stimulated conditions
* have a 12-lead ECG that is consistent with normal cardiac conduction and function
* have not used any tobacco products (eg, cigarettes, cigars, chewing tobacco, gum, or patch) for at least 6 months before first study drug administration

Exclusion Criteria:

* any personal or family history of epileptic seizures or convulsions
* have suffered from head trauma with loss of consciousness -have suffered from central nervous system infection
* have suffered from loss of consciousness of unknown origin
* drowning or sudden infant death syndrome in a first degree relative

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in vital signs and other parameters as a measure of safety and tolerability of tramadol | Baseline, Days 1 through 4
  Changes in clinical laboratory results, vital signs, psycopharmacologic status (Richmond Agitation-Sedation Scale (RASS), and physical examination.

SECONDARY OUTCOMES:
Change from baseline in time-matched electrocardiogram (ECG) measurements | Baseline, Day 1, Day 3 and Day 4
  ECG will detect abnormal changes from baseline in cardiac depolarization/repolarization.
Change from baseline in pharmacokinetic parameters of tramadol and M1 metabolite | Baseline, up to 72 hours after the 1st dose
  Determination of concentrations of tramadol and M1 metabolite pharmacokinetic parameters in venous plasma.
Incidence and type of adverse events | Baseline, till the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical trial, Study Director — Janssen Scientific Affairs, LLC
Locations (1):
- Overland Park, Kansas, United States